CLINICAL TRIAL: NCT03510377
Title: Effects of Aquatic Motor Intervention on Fall Risk, Hazard Perception for Pedestrians, Weekly Calendar Planning and Brain Activity During Elderly
Brief Title: Effects of Aquatic Intervention on Fall Risk, Hazard Perception, Calendar Planning and Brain Activity During Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Collaborators: The Science, Technology and Space Ministry, Israel (Unknown)
Responsible Party: Principal Investigator, Navah Ratzon, Professor, Occupational Therapist, Tel Aviv University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Michal Nissim
Record Dates: First submitted 2017-10-31; First posted 2018-04-27 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Aging; Falling; Pedestrian Accidents; Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Volunteers that will meet the inclusion criteria will be randomly divided to three intervention groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aquatic physical intervention (Experimental): Aquatic physical intervention: Ai-Chi
  Interventions: Other: Aquatic physical intervention; Other: On-land physical intervention; Other: Non physical intervention
- On-land physical intervention (Experimental): On-land physical intervention: Tai-Chi
  Interventions: Other: Aquatic physical intervention; Other: On-land physical intervention; Other: Non physical intervention
- Non physical intervention (Experimental): Non physical intervention: Guided imagery
  Interventions: Other: Aquatic physical intervention; Other: On-land physical intervention; Other: Non physical intervention

INTERVENTIONS:
Other: Aquatic physical intervention — For structured aquatic physical intervention group, the Ai-Chi method was selected. Ai-Chi is a simple aquatic exercise and relaxation method that uses a combination of deep breathing and slow movements of the arms, legs and torso in continual flowing patterns. The Ai-Chi intervention will occur in an hydrotherapy pool (34C).
Other: On-land physical intervention — For controlled comparison of the structured physical intervention group the Tai-Chi method was selected (the same movements as the Ai-Chi). The Tai-Chi intervention will occur in a room.
Other: Non physical intervention — The people who will be part of the non physical intervention will practice guided imagery of the Ai-Chi method. The guided imagery intervention will occur in a room.

SUMMARY:
Normal aging is associated with balance, mobility and executive functions decline that increase fall risk and influence Activity of Daily Living (ADL) and Instrumental ADL (IADL) functions such as safe road-crossing, planning and organizing everyday activities. Changes in cerebellar functional plasticity may mediate between the decline in balance, mobility and executive functions during elderly. Fortunately, mounting evidence suggests that physical activity is beneficial for decreasing aging effects and optimize brain structure and function. According to the dynamic systems theory, the environment in which the physical activity occurs influences the results of the activity. We propose an aquatic physical intervention program as a tool to decrease aging effects that in turn might lower fall risk, increase safety of road-crossing and improve planning and organizing everyday activities among community-dwelling older individuals.

DETAILED DESCRIPTION:
The percentage of elderly individuals (65+) in the society of Israel is 10.6%. As life-span increases, this percentage is expected to reach 15% in 2035. According to the Central Bureau of Statistics of Israel regarding the injuries and fatalities of road users, about 14% of the injuries and about 42% of the fatalities are pedestrians. Older pedestrians are about 22% of the pedestrians, twice their part in the population. Ageing effects on balance, mobility and executive functions (especially working memory and inhibitory control) might partially explain these statistics.

Changes in cerebellar functional plasticity may mediate between the decline in balance, mobility and some executive functions during elderly. Studies have shown age-related decrease in structural morphology and function of the cerebellum. The traditional functions of the cerebellum mainly include involvement in the coordination of motor movements, maintenance of balance, and motor learning. Interestingly, studies have found that cerebellar alpha power has an important role in voluntary movement, as well as in higher non-motor cognitive functions such as working memory. Cerebellar activation during working memory task may reﬂect the automated simulation of cognitive operations.

Various forms of physical interventions were found beneficial to promote balance, mobility and executive function of working memory and inhibitory control performances and optimize brain structure and function during elderly. The environment in which the physical intervention occurs is important. Therefore, changing the environment of intervention from on-land to aquatic may result in changing of cerebellar activity, thereby influence on balance, mobility, working memory and inhibitory control abilities proven to be functions connected to the cerebellum.

Due to the characteristics of water (such as density and viscosity), an immersed individual is exposed to physical forces (e.g. specific gravity, thermodynamics and the meta-centric effect) that do not exist on land. Immersion improves balancing abilities by increasing the proprioceptive input to the immersed body. Sensory feedback is increased by promoting a sense of body awareness, as resistance to movement through water is greater than resistance to movement through air. In support of this view, a recent Magnetoencephalography (MEG) study among adults has shown improved verbal working memory ability following one month of intensive aquatic physical intervention. Improved verbal working memory was positively correlated with increased right cerebellar alpha power. In the purpose study we examine the effects of physical intervention in different environments on balance, mobility, working memory and inhibitory control abilities and brain activity in order to decrease aging effects that in turn might lower fall risk, increase safety of road users and improve planning and organizing everyday activities among community-dwelling older individuals.

ELIGIBILITY:
Inclusion Criteria:

* Score less than 10 on the Geriatric Depression Scale
* Score above 24 in the Mini Mental State Examination

Exclusion Criteria:

* A medical history of neurological, orthopedic and/or psychiatric conditions with permanent impairments, or using drugs that according to the guidelines of the pharmaceutical company may cause dizziness
* Absence of longer than one week from the intervention

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Change in the Tinetti balance, gait and fall risk test | Change from Baseline to 1.5 months of intervention and to 3 months of intervention
  This test is a standardized evaluation of balance and mobility designed to determine risk for falls during elderly. It has a very good inter-rater reliability and sensitivity. The gait testing included initiation of gait, step height, step length, step symmetry, step continuity, path deviation, trunk stability, walk stance, and turning while walking. Each item scored 1 if normal or 0 if abnormal. The balance testing included sitting balance, arising from chair, immediate standing, standing balance, balance with eyes closed, turning balance, neck turning, back extension, one-leg standing, push test, reaching up, bending down, and sitting down. Each item scored 1 (normal) or 0 (abnormal). Tinetti scores for risk of falls: ≤18 points=high risk; 19-23 points=moderate risk; ≥24 points =low risk.
Change in digit span forward and backward tests | Change from Baseline to 1.5 months of intervention and to 3 months of intervention
  During the task a sequence of digits is read by the experimenter at a rate of 1/second, and participants is asked to recall the digits in forward or backward order immediately after hearing them. The task starting with a sequence of two digits, the number of digits per sequence will increase by one if a participant successfully recall a given sequence length twice. Testing will end when the participant makes errors on two successive trials of a given length. Performance will express as the number of sequences successfully recall.
Change in Corsi block forward and backward tests | Change from Baseline to 1.5 months of intervention and to 3 months of intervention
  During the tasks the subject watches the tester touch a series of blocks (one block per second), then the subject is to touch the blocks in the same order or backward. The task starting with one block, the blocks per sequence will increase by one if a participant successfully recall a given sequence length twice. Testing will end when the participant makes errors on two successive trials of a given length. Performance will express as the number of sequences successfully recall.
Change in the Stroop test | Change from Baseline to 1.5 months of intervention and to 3 months of intervention
  This task measures inhibitory control which is one of the core elements of executive functions. The task involves showing words that are the names of colors. The letters making up each word are printed in a color of ink different from the color name the word represents. The participant is asked to quickly respond with the color ink he sees, and inhibit the printed word. Performance will express the time (in seconds) it takes to finish the task and accuracy.
Change in the weekly calendar planning activity test | Change from Baseline to 3 months of intervention
  This tool was designed to be useful across a variety of populations that exhibit difficulties in executive functioning. It provides a broad analysis of how a person manages and copes with a complex and cognitively challenging activity. In addition to including a weekly schedule, the assessment features client profiles on error analysis, visual performance, awareness of task difficulty, and pre/post comparisons. The Weekly Calendar Planning Activity has three levels of difficulty, from Level 1, the easiest, in which appointments are preordered, to Level 3, the most difficult, in which appointments are randomly ordered in paragraph form. We will use Level 2 for this study, In Level 2 the participant is presented with a list of appointments in random order they have to schedule during 1 week by filling in a paper calendar.
Change in the hazard perception test for pedestrians | Change from Baseline to 3 months of intervention
  This computerized test was aimed to test and train pedestrians to safe cross walking and detect on road hazards as soon as possible.
Change in brain activity during n-back test | Change from Baseline to 3 months of intervention
  Functional Magnetic Resonance Imaging (fMRI) is a non-invasive technology. The fMRI paradigm consists of 5 minutes resting-state and an N-back task. We will use the 3.0 Tesla Siemens Prisma MRI Scanner located in Tel-Aviv University.

CONTACTS AND LOCATIONS:
Overall Officials: Navah Ratzon, Prof., Principal Investigator — Tal Aviv University
Locations (1):
- Sackler Faculty of Medicine, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nissim M, Livny A, Barmatz C, Tsarfaty G, Berner Y, Sacher Y, Giron J, Ratzon NZ. Effects of aquatic physical intervention on fall risk, working memory and hazard-perception as pedestrians in older people: a pilot trial. BMC Geriatr. 2020 Feb 19;20(1):74. doi: 10.1186/s12877-020-1477-4. PMID 32075583